CLINICAL TRIAL: NCT00271635
Title: Phase 2 Study of Ascorbic Acid Treatment in Charcot-Marie-Tooth Type 1A
Brief Title: Ascorbic Acid Treatment in CMT1A Trial (AATIC)
Acronym: AATIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: C. Verhamme, MD, Academic Medical Center, university of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04/320
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Charcot-Marie-Tooth Disease; Hereditary Motor and Sensory Neuropathies
Keywords: Charcot-Marie-Tooth Disease; Hereditary Motor and Sensory Neuropathies; Ascorbic Acid; Vitamin C
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Hereditary Sensory and Motor Neuropathy | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ascorbic acid
  Interventions: Drug: ascorbic acid
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo 4 capsules b.i.d. during 1 year
  Arms: 2
Drug: ascorbic acid — Ascorbic acid 1000 mg (4 capsules of 250 mg) b.i.d. during 1 year
  Other Names: Vitamin C
  Arms: 1

SUMMARY:
Charcot-Marie-Tooth type IA (CMT1A) is the most prevalent hereditary peripheral neuropathy. Demyelination of peripheral nerves is the hallmark of CMT1A. Ascorbic acid has been shown to have a favorable influence on myelination in in vitro studies and in a mouse model for CMT1A. We will study the efficacy and safety of ascorbic acid treatment in young patients with CMT1A.

DETAILED DESCRIPTION:
Charcot-Marie-Tooth type 1A (CMT1A), or hereditary motor and sensory neuropathy type Ia (HMSN Ia), is an autosomal dominant disease, most often caused by a 1.5 Mb duplication of chromosome 17, giving rise to three copies of the peripheral myelin protein 22 gene (PMP22). Mutations in this gene rarely cause CMT1A. It is a primarily demyelinating neuropathy, as has been shown in nerve conduction studies and in histopathological investigations. The conduction velocities of peripheral nerves are already slowed at the age of five years. Longitudinal data show that these conduction velocities do not change during life, indicating that the degree of demyelination is rather constant during life.

CMT1A is characterized clinically by distal muscle weakness and wasting, legs more than arms, impaired distal sensation, and reduced or absent reflexes. Moreover, foot and hand deformities are often encountered. In childhood, disease progression has been shown. In adults, there are indications for disease progression, but properly conducted longitudinal studies are awaited. Cross-sectional studies show that disease severity in adults is variable: a group of CMT1A patients is asymptomatic (5-10%), whereas other patients are wheelchair dependent (5-10%), still most have the classical CMT phenotype. Therapy is symptomatic and aims at maintaining functional possibilities and learning compensation mechanisms. There is no medication available that stabilizes or improves the clinical signs and symptoms.

Ascorbic acid is needed in in vitro studies for proper myelination of axons (in cultures containing serum). Recently, in a mouse model for CMT1A it has been shown that ascorbic acid improves the CMT1A phenotype. Mice (2-4 months old) treated with ascorbic acid once a week during three months showed an increase in the percentage of myelinating nerve fibers and showed better results in locomotor tests.

In this phase 2 study we will study the efficacy and safety of ascorbic acid in young patients with CMT1A. We will investigate whether ascorbic acid induces remyelination by measuring the nerve conduction of a peripheral nerve during a one year study period. CMT1A patients aged 12 years or older may cooperate sufficiently in nerve conduction studies. We include young patients, as clinical signs and symptoms especially develop relatively early in life. These signs and symptoms are due to axonal dysfunction, secondary to the demyelination. This is why we will investigate additionally whether there is an effect of ascorbic acid treatment on axonal function, strength and disabilities.

ELIGIBILITY:
Inclusion Criteria:

* DNA-proven CMT1A patients
* Age 12-25 years
* CMT 1A patients with symptomatology defined as muscle weakness in at least foot dorsiflexion

Exclusion Criteria:

Due to possible influence on severity of the neuropathy:

* Known other disease that may cause a neuropathy, that may decrease mobility, or that may lead to severe disability or death in a short time
* Medication that may cause a neuropathy
* Chronic alcohol abuse

Due to study medication (ascorbic acid):

* Regular use of vitamin C
* Clinical or echographic signs of nephrolithiasis
* Reduced glomerular filtration rate
* Iron overload
* No regular dental control at the dentist
* Pregnancy or active pregnancy wish for women

Due to study design and primary outcome:

* Not signing the informed consent
* Psychiatric co-morbidity which may influence compliance
* Not being comfortable during nerve conduction studies of the median nerve
* A too small CMAP amplitude of the abductor pollicis brevis muscle for a proper determination of the nerve conduction velocity of the median nerve

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in motor nerve conduction velocity of the median nerve after 1 year | 1 year

SECONDARY OUTCOMES:
Change in minimal F response latency of the median nerve after 1 year | 1 year
Changes in compound muscle action potential amplitude and area after 1 year | 1 year
Change in motor unit number estimation of the abductor pollicis brevis muscle after 1 year | 1 year
Changes in handgrip strength, strength of armflexors, foot dorsiflexors, knee extensors and hip flexors after 1 year | 1 year
Change in overall disability sum score after 1 year | 1 year
Change in AMC Linear Disability Scale score after 1 year | 1 year
Evaluation of serum ascorbic acid concentrations during 1 year | 1 year
Evaluation of side effects during 1 year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: C. Verhamme, MD, Principal Investigator — Department of Neurology, Academic Medical Center, University of Amsterdam; M. Vermeulen, MD, PhD, Principal Investigator — Department of Neurology, Academic Medical Center, University of Amsterdam; F. Baas, MD, PhD, Principal Investigator — Department of Neurology, Academic Medical Center, University of Amsterdam; R. de Haan, MD, PhD, Principal Investigator — Department of Neurology, Academic Medical Center, University of Amsterdam; M. de Visser, MD, PhD, Principal Investigator — Department of Neurology, Academic Medical Center, University of Amsterdam; I. N van Schaik, MD, PhD, Principal Investigator — Department of Neurology, Academic Medical Center, University of Amsterdam
Locations (1):
- Department of Neurology Academic Medical Center University of Amsterdam, Amsterdam, P.O.Box 22660, Netherlands

REFERENCES:
- [Background] Passage E, Norreel JC, Noack-Fraissignes P, Sanguedolce V, Pizant J, Thirion X, Robaglia-Schlupp A, Pellissier JF, Fontes M. Ascorbic acid treatment corrects the phenotype of a mouse model of Charcot-Marie-Tooth disease. Nat Med. 2004 Apr;10(4):396-401. doi: 10.1038/nm1023. Epub 2004 Mar 21. PMID 15034573
- [Background] Verhamme C, van Schaik IN, Koelman JH, de Haan RJ, Vermeulen M, de Visser M. Clinical disease severity and axonal dysfunction in hereditary motor and sensory neuropathy Ia. J Neurol. 2004 Dec;251(12):1491-7. doi: 10.1007/s00415-004-0578-x. PMID 15645349
- [Derived] Verhamme C, de Haan RJ, Vermeulen M, Baas F, de Visser M, van Schaik IN. Oral high dose ascorbic acid treatment for one year in young CMT1A patients: a randomised, double-blind, placebo-controlled phase II trial. BMC Med. 2009 Nov 12;7:70. doi: 10.1186/1741-7015-7-70. PMID 19909499